CLINICAL TRIAL: NCT05480605
Title: Characterizing Occupational Therapy Intervention for Children With Autism Spectrum
Brief Title: Characterizing Occupational Therapy Intervention for Children With Autism Spectrum Disorders
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: American Occupational Therapy Foundation (Other); Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Jewel Crasta, Assistant Professor, Ohio State University
Other Study IDs: 2021H0140
Record Dates: First submitted 2022-04-18; First posted 2022-07-29 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Occupational Therapy; Engagement; Autism Spectrum Disorders; EEG/ERP
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Occupational Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental Group: Children with autism ages 6-13
  Interventions: Behavioral: Occupational Therapy

INTERVENTIONS:
Behavioral: Occupational Therapy — Children with autism will receive 6 - 8 weeks of regularly scheduled occupational therapy at Nationwide Children's Hospital outpatient centers. The intervention consists of one-hour weekly sessions with a licensed occupational therapist.

SUMMARY:
This pilot study aims to identify behavioral and neural measures of sensory processing and attention associated with routine occupational therapy intervention for children with autism spectrum disorders. Specifically, the investigator will examine the impact of a child's level of engagement during therapy using standardized behavioral and electroencephalography (EEG) measures of sensory processing.

DETAILED DESCRIPTION:
Occupational therapy is one of the most frequently requested and highly utilized interventions for children with autism spectrum disorders (autism) and therapists have consistently reported using the sensory integration framework as a dominant theory guiding practice. A key component of sensory integration theory is the child's active engagement during therapy, which is assumed to improve neural function, behavior, and participation. However, no studies have examined the neural mechanisms associated with occupational therapy interventions among children with autism.

This pilot feasibility study will examine behavioral and electroencephalography (EEG) measures of attention and sensory processing before and following 6-8 weeks of routine occupational therapy at community outpatient centers among 30 children with autism aged 6 - 13 years. The primary aim is to determine the feasibility, sensitivity, and validity of EEG measures of auditory processing as a response biomarker following routine occupational therapy intervention. Another aim is to examine the contribution of a child's engagement during therapy as a key predictor of change using behavioral and EEG outcome measures. The occupational therapy intervention consists of one-hour weekly sessions of usual care at Nationwide Children's Hospital outpatient centers.

Results from this grant will provide valuable proof-of-concept data establishing engagement during therapy as an active ingredient in occupational therapy intervention using neurophysiological and behavioral measures. These results will also establish the validity of EEG measures as sensitive to a child's level of engagement and neuroplastic changes following occupational therapy intervention.

ELIGIBILITY:
Inclusion Criteria:

For children with autism:

* a medical diagnosis of Autism
* between 8 - 13 years
* must be verbal
* have normal or corrected vision/hearing
* enrollment in the 8-week OT treatment plan with a therapist enrolled in the study.

For typically developing children:

• No history of neurological injuries, disabilities, and family history of mental health disorders on parent report

Exclusion Criteria:

* history of a definitive neurologic disorder including seizures (except for uncomplicated brief febrile seizures), tumor, severe head injury, stroke, lesion, or disease
* presence of a severe chronic medical disorder
* presence of a major visual impairment
* history of alcohol/substance abuse or dependency.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children ages 6-13 years diagnosed with Autism with an IQ > 65, and age-matched typically developing children.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
EEG: Changes in Sensory Gating event-related potential (ERP) measures. | 8 weeks
  Amplitudes and latencies of the P50 and N1 ERP components from the sensory gating paradigm. The P50 component presents as a positive deflection that occurs around 40-80 milliseconds (ms) after click onset and the N1 represents a negative deflection occurring around 100 ms. Gating will be assessed using difference scores wherein the amplitude of click 2 is subtracted from the amplitude of click 1.
EEG: Changes in Sensory Gating neural oscillations | 8 weeks
  Evoked and phase-locked Beta power (13-18 Hz) and Gamma power (30-50 Hz) following click onset will be examined.
EEG: Changes in Sensory Registration event-related potential (ERP) | 8 weeks
  The Sensory Registration paradigm consists of four tones of different frequencies and intensities. Amplitude and latency of the P1, N1, P2, N2, and P3 ERP measures following the four tones of the sensory registration paradigm will be examined.
Changes in behavioral measure of Social Responsiveness | 8 weeks
  The Sensory Responsiveness scale - 2 (SRS-2) is a standardized parent-report measure and will be used to measure social responsiveness.
Changes in behavioral measure of Sensory Processing | 8 weeks
  The Sensory Profile - 2 (SP2) is a standardized parent-report measure and will be used to measure sensory processing.
Changes in behavioral measure of Attention | 8 weeks
  The Test of Everyday Attention for Children 2 (TEA-Ch2) will be used to measure attention. The TEACh2 is a standardized performance-based measure.

SECONDARY OUTCOMES:
Changes in Behavioral measures of executive functioning | 8 weeks
  The Behavior Rating Inventory of Executive Function-2 (BRIEF-2) is a standardized parent-report measure of executive functioning.
Changes in behavioral measure of Adaptive behavior | 8 weeks
  The Vineland Adaptive Behavior Scales-3 (VABS-3) is a standardized parent-report measure of adaptive behavior and is widely used in autism research.
Changes in behavioral measures of Anxiety | 8 weeks
  The Children's Anxiety Scale (SCAS) is a parent-report measure of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Jewel Crasta, PhD., OTR/L, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Nationwide Children's Hospital, Columbus, Ohio
  - McCampbell Hall, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be released at the end of the study and accessible upon request.
Access Criteria: IPD will be accessible upon request to the study PI.

REFERENCES:
- [Background] Case-Smith J, Weaver LL, Fristad MA. A systematic review of sensory processing interventions for children with autism spectrum disorders. Autism. 2015 Feb;19(2):133-48. doi: 10.1177/1362361313517762. Epub 2014 Jan 29. PMID 24477447
- [Background] Crasta, J. E. (2018). Behavioral and neural sensory processing in young adults with autism spectrum disorder. American Journal of Occupational Therapy, 72(4_Supplement_1), 7211505081p1. https://doi.org/10.5014/ajot.2018.72S1-PO1012
- [Background] Dawson G, Jones EJ, Merkle K, Venema K, Lowy R, Faja S, Kamara D, Murias M, Greenson J, Winter J, Smith M, Rogers SJ, Webb SJ. Early behavioral intervention is associated with normalized brain activity in young children with autism. J Am Acad Child Adolesc Psychiatry. 2012 Nov;51(11):1150-9. doi: 10.1016/j.jaac.2012.08.018. PMID 23101741
- [Background] LaGasse AB, Manning RCB, Crasta JE, Gavin WJ, Davies PL. Assessing the Impact of Music Therapy on Sensory Gating and Attention in Children With Autism: A Pilot and Feasibility Study. J Music Ther. 2019 Aug 13;56(3):287-314. doi: 10.1093/jmt/thz008. PMID 31225588
- [Background] Miller LJ, Anzalone ME, Lane SJ, Cermak SA, Osten ET. Concept evolution in sensory integration: a proposed nosology for diagnosis. Am J Occup Ther. 2007 Mar-Apr;61(2):135-40. doi: 10.5014/ajot.61.2.135. No abstract available. PMID 17436834
- [Background] Crasta JE, Gavin WJ, Davies PL. Expanding our understanding of sensory gating in children with autism spectrum disorders. Clin Neurophysiol. 2021 Jan;132(1):180-190. doi: 10.1016/j.clinph.2020.09.020. Epub 2020 Oct 16. PMID 33310588